CLINICAL TRIAL: NCT04737967
Title: The Potential Protective Role of Venlafaxine Versus Memantine in Paclitaxel Induced Peripheral Neuropathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mendel AI (Industry)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, G Fadl, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIPN101
Record Dates: First submitted 2021-01-30; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Oncology Pain; Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: conditions — Cancer Pain | interventions — Venlafaxine Hydrochloride; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venlafaxine Treated Arm (Experimental)
  Interventions: Drug: Venlafaxine
- Memantine Treated Arm (Experimental)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Venlafaxine — Patients will receive will receive Venlafaxine extended release (37.5 mg) tablets once daily(Zimmerman et al., 2016)
  Arms: Venlafaxine Treated Arm
Drug: Memantine — Patients will receive memantine (10 mg) once daily (Morel et al., 2016)
  Arms: Memantine Treated Arm

SUMMARY:
This is a double blinded two-arm randomized case-only interventional trial. A total of 60 patients who are to receive Paclitaxel to be included and allocated in two groups. The protocol is to be reviewed by the Research Ethics Committee of Faculty of Medicine Cairo University.

All procedure will be done in Kasr El-Einy Center of Radiation Oncology and Nuclear Medicine.

The first arm (Venlafaxine group) will receive Venlafaxine extended release (37.5 mg) tablets (Zimmerman et al., 2016).

The second arm (Memantine group) will receive memantine 10 mg once daily (Morel et al., 2016)

ELIGIBILITY:
Inclusion Criteria:

1. All patients, 18 years of age or older, with a cancer treated with Paclitaxel
2. Patients must have a life expectancy of at least 24 weeks.
3. Patients must sign an informed consent.
4. Patients may have a grade 0 (chemotherapy naive) or 1 neuropathy (history of prior chemotherapy) prior to entry.
5. Patient matching high risk on the CIPN risk stratification scoring system

Exclusion Criteria:

1. Patients with symptomatic brain metastases.
2. Pregnant women or nursing mothers. Patients of child bearing potential must use adequate contraception.
3. Patients may receive no other concurrent complementary medicines during this study.
4. Patients with neuropathy induced diabetes.
5. Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in average daily pain intensity | 6 weeks
  Change in average daily pain intensity as measured by the Brief Pain Inventory- Short Form (BPI-SF). Absolute change in the average daily pain intensity as measured by the Brief Pain Inventory- Short Form (BPI-SF) from baseline to the end of 6 weeks measured by item # 5 of Brief Pain Inventory Score (BPI-SF). The BPI assesses pain at its "worst," "least," "average," and "now" (current pain).
Electrophysiological studies | 6 weeks
  nerve conduction velocity at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Cairo University - Kasr El-Einy Center of Radiation Oncology and Nuclear Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No